CLINICAL TRIAL: NCT02201654
Title: Stylet Versus no Stylet in Endobronchial Ultrasound Transbronchial Aspiration (EBUS-TBNA)
Brief Title: Stylet vs No Stylet During EBUS TBNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NA_00093452
Record Dates: First submitted 2014-06-05; First posted 2014-07-28 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

ARMS (1):
- EBUS patients (Other): All patients in our study are in the same arm, as each patient serves as their own internal control. More specifically, each enrolled patient will receive both traditional EBUS (with the usage of stylet) and experimental EBUS (EBUS without a stylet) at each lymph node that is included in the experimental analysis.
  Interventions: Other: EBUS without stylet

INTERVENTIONS:
Other: EBUS without stylet — the patient will receive both conventional ebus with the stylet and experimental ebus (without the stylet). The two techniques will then be compared to each other on a per lymph node basis.

SUMMARY:
This research study compares two ways to biopsy lymph nodes in the chest using endobronchial ultrasound-guided transbronchial needle aspiration" (EBUS-TNBA). During a EBUS-TBNA procedure, the patient is sedated, and a flexible camera and ultrasound probe is inserted through the mouth into the large airways of the chest, allowing us to see (via ultrasound) and biopsy the lymph nodes in the chest.

The purpose of this research study is to determine if the EBUS-TBNA procedure can be made simpler. In today's practice, the biopsy needle has two parts, 1) the needle itself and 2) an inner stylet that runs through the middle of the needle. Because many other biopsy needles (such as the needles used in breast biopsy and different types of lung biopsy needles) do not use an inner stylet, the investigators do not think the use of a stylet is necessary. If this step can be safely eliminated without decreasing the effectiveness of the procedure, this could shorten the procedure (saving time). This study is deigned to formally test the hypothesis that a stylet is not necessary in EBUS-TBNA.

ELIGIBILITY:
Inclusion Criteria:

* All patients >18 years old and capable of informed consent refereed for EBUS-TBNA at our institution.

Exclusion Criteria:

* Standard contraindications to EBUS (coagulopathy, anti-platlet/anti-coagulant use, clinical instability)
* Pregnant women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic agreement (percentage of samples that have the same diagnosis) | At time of biopsy
  The main outcome is the agreement (concordance) between the pathological diagnosis obtained by preforming EBUS with a stylet with EBUS without a stylet. Each patient will receive both techniques on each lymph node. We will then compare the diagnostic reached by each technique, and calculate the percentage of the time these techniques result in the same diagnosis.

SECONDARY OUTCOMES:
Pneumothorax rate (percentage of procedures that result in a pneumothorax) | 1 week post-procedure
  Complications related to EBUS-TBNA are very rare, and are not anticipated to be higher due to enrollment in this study. We will track complications such as excessive bleeding, pneumothorax, and unanticipated admission to the hospital
Bleeding rate (% of procedures that have significant bleeding) | 1 week post-procedure
  Complications related to EBUS-TBNA are very rare, and are not anticipated to be higher due to enrollment in this study. We will track complications such as excessive bleeding, pneumothorax, and unanticipated admission to the hospital
Hospital Admission (% of procedures that result in unanticipated admission to the hospital) | 1 week post-procedure
  Complications related to EBUS-TBNA are very rare, and are not anticipated to be higher due to enrollment in this study. We will track complications such as excessive bleeding, pneumothorax, and unanticipated admission to the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States